CLINICAL TRIAL: NCT06837623
Title: The Role of Colchicine as Anti-Inflammatory Treatment in Patients With HFpEF: A Prospective Study
Brief Title: Role of Colchicine as Anti-Inflammatory Therapy in HFpEF
Acronym: CO-HFpEF
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaima Mohammed Zeyad, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ms-220-2024
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; Colchicine
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group/Arm (Experimental): Eligible HFpEF patients with a body weight of ≥70 kg will receive colchicine 0.5 mg twice daily, while those weighing <70 kg will receive 0.5 mg once daily, in addition to usual care for 12 weeks.
  Interventions: Drug: Colchicine Tablets

INTERVENTIONS:
Drug: Colchicine Tablets — Oral colchicine tablets. The dosing regimen is as follows:
  * Patients weighing >70 kg: 0.5 mg twice daily (BID)
  * Patients weighing ≤70 kg: 0.5 mg once daily (OD) Administered for 3 months
  Other Names: Colchicine

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a condition associated with high morbidity and mortality. Chronic low-grade inflammation plays a key role in its progression, yet few treatments specifically target this pathway.

This clinical trial aims to evaluate the effectiveness of colchicine, a well-tolerated anti-inflammatory drug, in reducing inflammation in HFpEF patients. The study will assess whether colchicine lowers levels of soluble ST2 (sST2), a biomarker linked to inflammation and cardiac stress in HFpEF.

Participants will take colchicine daily for three months, with blood samples collected at baseline and at the end of the study to measure changes in sST2 levels. The findings could provide new insights into the potential role of colchicine as a treatment for HFpEF.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a complex condition associated with high morbidity and mortality. While its exact causes remain unclear, low-grade systemic inflammation plays a key role by promoting myocardial fibrosis and increasing heart muscle stiffness. Despite this, anti-inflammatory treatments for HFpEF remain largely unexplored.

Colchicine is a well-established anti-inflammatory drug that blocks key inflammatory pathways, including inflammasome activation and the release of interleukin-1 (IL-1). It has demonstrated cardiovascular benefits in trials such as COLCOT and LoDoCo2, significantly reducing the risk of heart-related events in coronary artery disease. However, its effects in HFpEF patients are not yet known.

Two important biomarkers-soluble suppression of tumorigenicity 2 (sST2) and high-sensitivity C-reactive protein (hsCRP)-are strongly linked to worse outcomes in HFpEF. Elevated sST2 reflects increased fibrosis and cardiac stress, while high hsCRP indicates systemic inflammation. Both markers are associated with more severe symptoms and a higher risk of complications. Additionally, the 6-minute walk test (6MWT) is a widely used measure of physical function and exercise capacity in heart failure patients.

This single-center, prospective clinical trial aims to evaluate the effects of colchicine in HFpEF patients with elevated inflammation. Participants will receive colchicine for three months, with assessments of sST2, hsCRP, and 6MWT performance before and after treatment. Findings from this study may provide valuable insights into whether colchicine can reduce inflammation and improve functional capacity in HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age, males and females.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
* Symptoms and/or signs of heart failure.
* H2FPEF score ≥ 6 points or HFA-PEFF score ≥ 5 points.
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≥125 pg/mL at baseline (patients with atrial fibrillation at baseline NT-proBNP ≥365 pg/mL), or objective evidence of systemic or pulmonary congestion.
* Stable medical therapy within the last 1 month.

Exclusion Criteria:

* Patients requiring colchicine for other conditions or with a history of colchicine intolerance or hypersensitivity.
* Active or chronic inflammatory diseases or infection.
* Presence of active solid tumors or hematological malignancies.
* Estimated glomerular filtration rate (eGFR) <35 mL/min/1.73 m².
* Severe liver disease includes Child-Pugh class B or C, cirrhosis, or chronic active hepatitis.
* Concurrent use of strong CYP3A4 or P-glycoprotein inhibitors.
* Presence of blood dyscrasias.
* Recent major cardiovascular events or procedures within the last 3 months.
* Established diagnosis of pericardial disease, myocarditis, hypertrophic cardiomyopathy, and cardiac amyloidosis
* Significant valvular heart disease.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Soluble Suppression of Tumourigenicity 2 (sST2,ng/ml) | From baseline to 12 weeks post-treatment initiation
  Delta_circulating sST2

SECONDARY OUTCOMES:
Change in high-sensitivity C-reactive protein (hsCRP, mg/L) | From baseline to 12 weeks post-treatment initiation
  Delta_circulating_hsCRP
Change in 6 Minute Walk Test (6MWT,meters) | From baseline to 12 weeks post-treatment initiation
  Change in 6MWT distance

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Abdelhamid Abdel Aziz, Professor of Cardivascular M, Study Chair — Cairo University; Ahmed Kamal, MD in Cardiology, Principal Investigator — Cairo University; Nesrine M El Gharbawi, Prof of clin. & Chem Patho, Principal Investigator — Cairo University; Shaima M Zeyad, Cardiology Resident, Principal Investigator — Cairo University
Locations (1):
- Cairo University - Kasr Al-Ainy, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon reasonable request with a corresponding offer.